CLINICAL TRIAL: NCT04612803
Title: Observational Study of the Prevalence of Antihistamine Responsive Gastrointestinal Symptoms in Patients Diagnosed With Irritable Bowel Syndrome With Diarrhea
Brief Title: Prevalence of Antihistamine Responsive Irritable Bowel Syndrome With Diarrhea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, David Bernstein, Emeritus Professor of Medicine, University of Cincinnati
Other Study IDs: 2020-0193
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Irritable Bowel Syndrome; Dermatographism; Post-prandial Diarrhea
Keywords: IBS; irritable bowel syndrome; Dermatographism; post-prandial diarrhea; antihistamine
MeSH Terms: conditions — Irritable Bowel Syndrome; Familial dermographism | interventions — Histamine Antagonists

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- IBS-D + dermatographism: IBS-D patients with dermatographism. Cetirizine 10 mg and famotidine 20 mg will be dispensed to each patient, to be taken twice a day at 6-9AM one hour before eating breakfast and again at evening 12 hours after the morning dose for 30 days
  Interventions: Drug: Antihistamine

INTERVENTIONS:
Drug: Antihistamine — Cetirizine 10 mg and famotidine 20 mg will be dispensed to each patient, to be taken twice a day at 6-9AM one hour before eating breakfast and again at evening 12 hours after the morning dose for 30 days

SUMMARY:
Irritable bowel syndrome is a functional disorder of the gastrointestinal tract diagnosed with the Rome criteria. The Rome IV criteria are based on abdominal pain symptoms and stool habits including stool frequency and stool forms [1]. They define 3 main subtypes based on symptoms: 1) IBS with diarrhea; 2) IBS with constipation: and 3) mixed symptoms of constipation and diarrhea. The IBS with diarrhea (IBS-D) subtype has the highest prevalence. Currently, treatment of IBS-D includes antidiarrheals, bile acid sequestrants, antispasmodics, tricyclic antidepressants, and FODMAP diet. However, many patients are intolerant or unresponsive to the above treatments. Outside of IBS, chronic diarrhea affects about 5% of adults. We have described a syndrome in a subset of IBS patients presenting with post prandial diarrhea, flushing and dermatographia whose symptoms are prevented by pre-treatment with combined H1 and H2 antihistamines [2]. However, the prevalence of this syndrome among the IBS + D patients is not known nor have the clinical characteristics or predictors of antihistamine responsive IBS + D been defined.

DETAILED DESCRIPTION:
We have published a series of 5 patients with chronic post prandial diarrhea (PPD) that begins within 3 hours after eating, associated with dermatographia, responsive to antihistamines [2]. In these cases, no underlying causes were identified to explain PPD; diagnoses of food allergy, lactose intolerance, celiac disease, dumping syndromes, inflammatory bowel disease, systemic mastocytosis were excluded. Patients with the syndrome have prior histories of chronic urticaria and experience associated transient symptoms of flushing, headache, tachycardia, and abdominal bloating during PPD episodes.

This syndrome, except for our published report, have not been previously described in the medical literature. Patients with systemic mastocytosis and mast cell activation syndrome experience PPD but along with anaphylactic manifestations (e.g. wheezing, hypotension) and measurable mast cell biomarkers are identifiable in affected patients (i.e. serum mast cell tryptase or 24 hour urine methylhistamine, PGF2a). Therefore, it is important to characterize PPD responsive to antihistamines in a general GI patient population and to publish our findings. The impact on human health will be substantial; we found that these patients are undiagnosed and untreated for many years.

Our aim is to recruit 50-100 patients from the UC Health affiliated gastroenterology clinics with access UC health which has 300-500 potential subjects. We would need to recruit 10-20% percentage of these potential subjects. Kris Ramprasad MD, a faculty member in the Division of Gastroenterology, David Bernstein MD, a faculty member in the Division of Allergy and Rheumatology, allergy fellows and GI fellows will direct and implement subject screening and consenting.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Prior to Diagnosis of IBS + diarrhea based on ICD 10 codes with or without constipation unresponsive to prior treatments
* Moderate to severe symptom severity score (>175 points) based on IBS symptom severity scale
* Seeking evaluation by a health care professional
* Negative serologic celiac panel
* No response to lactose elimination diet by history
* Normal colonoscopy
* Able to complete symptoms diaries and global evaluations

Exclusion Criteria:

* Confirmed IgE dependent food allergy as a cause of the gastrointestinal symptoms.
* Lactose intolerance by history
* Celiac disease by serology
* Inflammatory bowel disease or colitis
* Bile acid diarrhea by history
* Post-surgical GI symptoms (e.g., dumping syndrome) by history
* No colonoscopy performed
* GI malabsorption
* Current pregnancy
* Current severe depression or history of psychosis
* Current treatment with tricyclic antidepressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a patient population of adults with chronic diarrhea that has been evaluated for the common causes and resulting with a diagnosis of exclusion: irritable bowel syndrome with diarrhea.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
IBS symptomy severity score | 135 days
  ≥50 point in reduction of symptoms with antihistamines based on the IBS symptom severity scale (IBS-SSS). This validated scale contains 5 questions that measures on a 100 point scale (for a total of 500 points) the severity of abdominal pain, frequency of abdominal pain, severity of abdominal distension, dissatisfaction with bowel habits, and interference with quality of life.

SECONDARY OUTCOMES:
IBS quality of life | 135 days
  ≥10 point improvement in Quality of Life (IBS-QOL) questionnaire and a "moderately improved" or "substantially improved" on the IBS global assessment of improvement (IBS-GAI) scale. The IBS-QOL is a 34-item questionnaire which assesses the degree to which IBS interferes with the patient's quality of life. The IBS-GAI asks one question that assesses the overall improvement in symptoms in the past 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: David Bernstein, MD, Principal Investigator — University of Cincinnati

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing individual participant data.

REFERENCES:
- [Background] Functional Gastrointestinal Disorders and the Rome IV process. In: Drossman DA, Chang L, Chey WD, Kellow J, Tack J, Whitehead WE, editors. Rome IV functional gastrointestinal disorders: disorders of gut-brain interaction.
- [Background] Hassoun Y, Stevenson MR, Bernstein DI. Idiopathic postprandial diarrhea responsive to antihistamines. Ann Allergy Asthma Immunol. 2019 Oct;123(4):407-409. doi: 10.1016/j.anai.2019.06.022. Epub 2019 Jul 3. No abstract available. PMID 31279076
- [Background] Mlynek A, Vieira dos Santos R, Ardelean E, Weller K, Magerl M, Church MK, Maurer M. A novel, simple, validated and reproducible instrument for assessing provocation threshold levels in patients with symptomatic dermographism. Clin Exp Dermatol. 2013 Jun;38(4):360-6; quiz 366. doi: 10.1111/ced.12107. PMID 23621090
- [Background] Patrick DL, Drossman DA, Frederick IO, DiCesare J, Puder KL. Quality of life in persons with irritable bowel syndrome: development and validation of a new measure. Dig Dis Sci. 1998 Feb;43(2):400-11. doi: 10.1023/a:1018831127942. PMID 9512138
- [Background] McHugh KR, Swamy GK, Hernandez AF. Engaging patients throughout the health system: A landscape analysis of cold-call policies and recommendations for future policy change. J Clin Transl Sci. 2018 Dec;2(6):384-392. doi: 10.1017/cts.2019.1. PMID 31402985
- [Background] Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther. 1997 Apr;11(2):395-402. doi: 10.1046/j.1365-2036.1997.142318000.x. PMID 9146781
- [Background] Passos MC, Lembo AJ, Conboy LA, Kaptchuk TJ, Kelly JM, Quilty MT, Kerr CE, Jacobson EE, Hu R, Friedlander E, Drossman DA. Adequate relief in a treatment trial with IBS patients: a prospective assessment. Am J Gastroenterol. 2009 Apr;104(4):912-9. doi: 10.1038/ajg.2009.13. Epub 2009 Mar 17. PMID 19293784
- [Background] Gordon S, Ameen V, Bagby B, Shahan B, Jhingran P, Carter E. Validation of irritable bowel syndrome Global Improvement Scale: an integrated symptom end point for assessing treatment efficacy. Dig Dis Sci. 2003 Jul;48(7):1317-23. doi: 10.1023/a:1024159226274. PMID 12870789
- [Background] B O'Neil, Some useful moment results in sampling problems. American Statistician Volume 69, Issue 4, 2014